CLINICAL TRIAL: NCT04123132
Title: Evaluation of Kinesophobia in Patients With Metabolic Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Erol Olcok Corum Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Dilek Eker Büyükşireci, Specialist doctor, Erol Olcok Corum Training and Research Hospital
Other Study IDs: 08090081DEB
Record Dates: First submitted 2019-10-09; First posted 2019-10-10 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Kinesiophobia; Metabolic Syndrome
Keywords: kinesiophobia; metabolic syndrome; exercise
MeSH Terms: conditions — Kinesiophobia; Metabolic Syndrome; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with metabolic syndrome
  Interventions: Other: Kinesiophobia
- Healthy controls

INTERVENTIONS:
Other: Kinesiophobia — The presence of kinesiofobia in patients with metabolic syndrome
  Groups: Patients with metabolic syndrome

SUMMARY:
Metabolic syndrome (MS) is a public health problem characterized by central obesity, increased blood pressure and triglyceride levels, decreased blood HDL levels and the presence of insulin resistance (1).Kinesiophobia is a fear of irrational movement that develops because of its belief in susceptibility to injury and is associated with low levels of physical activity. Considering that exercise improves metabolic processes in people with MS, we aimed to evaluate the presence of kinesophobia in patients with MS.

Patients aged 45-65 years diagnosed with metabolic syndrome and healthy controls will be included in the study. Patients with rheumatic and neurological diseases,history of trauma, gonarthrosis, lumbar disc hernia, previous fractures, fibromyalgia and those who have experienced pain for the last week will be excluded. The participants will be filled in the Short Form-36 (SF-36), the Hospital Anxiety and Depression Scale, and the Tampa Kinesiophobia Scale. 48 patients with MS and 48 healthy participants will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metabolic syndrome

Exclusion Criteria:

* Patients with rheumatic disease
* Patients with neurologic disease
* Patients with history of trauma
* Patients with gonartrosis
* Pateints with fibromialgia

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 45-65 years old men and female with metabolic syndrome and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2019-09-25 (Actual); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
Tampa Kinesiophobia Scale | 3 months
  People takes between 17-68 total a score. The score of the person shows high kinesiophobia on the scale

CONTACTS AND LOCATIONS:
Locations (1):
- Dilek Eker Büyükşireci, Çorum, Central Anatolia, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No